CLINICAL TRIAL: NCT05343026
Title: Efficacy of Hearing-aid Treatment on Sound Perception and Residual Hearing Preservation for Patients With Tinnitus and Co-existing Hearing Loss: a Randomized Controlled Trial
Brief Title: Efficacy of Hearing-aid Treatment for Patients With Tinnitus and Co-existing Hearing Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shan Sun
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Tinnitus, Subjective; Hearing Loss, High-Frequency
MeSH Terms: conditions — Tinnitus; Hearing Loss, High-Frequency | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA treatment group (Experimental): Participants in the treatment group are required to wear the HAs for at least 3 hours per day, with 24 days per month. Additionally, they will receive regular counseling and lifestyle education from their physicians.
  Interventions: Device: Hearing aids
- non-HA treatment group (No Intervention): Non-HA treatment group is a waiting list control group (WLC) in which participants will receive the intervention after the waiting period has passed. They will only receive regular counseling and lifestyle education from their physicians in this waiting period.

INTERVENTIONS:
Device: Hearing aids — As for screening the hearing and tinnitus testing, the measure typically comprises PTA, SRS, DPOAE, and several widely accepted standardized tinnitus questionnaires, including the THI for tinnitus severity and VAS for tinnitus loudness.
  Arms: HA treatment group

SUMMARY:
Considering the extent to which HAs play a role in sound perception and residual hearing preservation among patients with tinnitus and co-existing HL remains a lack of compelling extensive evidence, investigators designed this single-blind, 6-months randomized, controlled trial with two parallel groups. One is the HA treatment group, and the other is the waiting list control (WLC) group which receives no interventions during this period.

DETAILED DESCRIPTION:
In clinical practice, chronic subject tinnitus poses an important challenge. This condition can negatively affect an individual's emotional and functional well-being. In most cases, tinnitus is highly associated with hearing impairment, particularly in cases of high-frequency sensorineural hearing loss (SNHL). The occurrence of tinnitus in patients with HL is one of the most prevalent sensory disabilities, causing a deleterious effect on patients' lives. Nowadays, the mild to moderate SNHL can be effectively managed with a fitting hearing aid (HA) by providing sound amplification, and several findings suggest that the HA may also be helpful for people with tinnitus. Nevertheless, in terms of the effects of HA use for residual hearing protection for patients with tinnitus and co-existing hearing loss, inadequate attention is still paid by medical personnel, and relevant evidence remains preliminary at this point in time.

To assess the full extent of tinnitus patients, investigators need to carry out a series of tests, including hearing assessment and psychometric tests. Pure tone audiometry (PTA) and otoacoustic emission (OAE) tests are used to calculate the average hearing thresholds and the outer hair cell function, while the Tinnitus hazard Index (THI), the Visual Analogue Scale (VAS), the Hospital Anxiety and the Depression Scale (HADs) and the Athens Insomnia Scale-8 (AIS-8) questionnaires were for patients' psychology status.

Investigators hypothesize that in patients with tinnitus and hearing loss, HA intervention results in better conditions of tinnitus and lower hearing threshold reduction. Here investigators planned to enroll patients into two groups, the HA and non-HA (served as the control) intervention patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged older than 18 years old and less than 70 years;
2. Chronic (>6 months) subjective tinnitus, unilateral or bilateral;
3. Diagnosed with a high-frequency SNHL;
4. Be available for six months after starting the study to complete the follow-up questionnaires;
5. Readiness to participate in the study and sign the informed consent.
6. Be covered by public health insurance and eligible for reimbursement.

Exclusion Criteria:

1. Objective tinnitus;
2. Conductive HL;
3. Unstable medical history that limits participation;
4. Undergoing any other concurrent treatments on tinnitus or HL;
5. Having used HAs in the past 1 year;
6. Unwilling or unable to use HAs daily;
7. Alcohol or drug abuse;
8. Unable to read or write.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
tinnitus handicap inventory (THI) | 3 months from baseline
  The THI is a self-administered test, including 25 questions with grades four categories of tinnitus severity: slight corresponding to a score of 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus.
tinnitus handicap inventory (THI) | 6 months from baseline
  The THI is a self-administered test, including 25 questions with grades four categories of tinnitus severity: slight corresponding to a score of 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus.

SECONDARY OUTCOMES:
speech recognition score (SRS) test | 3 months from baseline
  The list consists of 25 monosyllabic words, and each word is rated on a 4-point scale with a total score of 100. A higher score indicates a better level of auditory comprehension and speech recognition.
speech recognition score (SRS) test | 6 months from baseline
  The list consists of 25 monosyllabic words, and each word is rated on a 4-point scale with a total score of 100. A higher score indicates a better level of auditory comprehension and speech recognition.
pure tone audiometry (PTA) | 3 months from baseline
  PTA is performed to calculate the average hearing thresholds obtained at multiple frequencies in dB hearing level.
pure tone audiometry (PTA) | 6 months from baseline
  PTA is performed to calculate the average hearing thresholds obtained at multiple frequencies in dB hearing level.
otoacoustic emission (OAE) | 3 months from baseline
  OAE test could help evaluate the mechanism of tinnitus since it determines whether or not the outer hair cells are overexcited or damaged.
otoacoustic emission (OAE) | 6 months from baseline
  OAE test could help evaluate the mechanism of tinnitus since it determines whether or not the outer hair cells are overexcited or damaged.
the Hospital Anxiety and Depression Scale (HADs) | 3 months from baseline
  The HADs consist of 14 items which are equally divided into two dimensions: a depression sub-scale (HADs-D) and an anxiety sub-scale (HADs-A). The grades are valued by scoring: negative (0-7), positive (8-21).
the Hospital Anxiety and Depression Scale (HADs) | 6 months from baseline
  The HADs consist of 14 items which are equally divided into two dimensions: a depression sub-scale (HADs-D) and an anxiety sub-scale (HADs-A). The grades are valued by scoring: negative (0-7), positive (8-21).
the Athens Insomnia Scale-8 (AIS-8) | 3 months from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).
the Athens Insomnia Scale-8 (AIS-8) | 6 months from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).

CONTACTS AND LOCATIONS:
Overall Officials: Shan Sun, Principal Investigator — Eye and ENT Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li P, Tang D, Wu Y, Yin Y, Sun S. Efficacy of hearing aid treatment on sound perception and residual hearing preservation in patients with tinnitus and coexisting hearing loss: study protocol for a randomized controlled trial. Trials. 2022 Dec 27;23(1):1049. doi: 10.1186/s13063-022-07014-0. PMID 36575531